CLINICAL TRIAL: NCT00002268
Title: A Randomized, Phase I/II Trial to Assess the Safety and Antiviral Effects of Escalating Doses of A Human Anti-Cytomegalovirus Monoclonal Antibody (SDZ MSL-109) in Patients With the Acquired Immunodeficiency Syndrome and CMV Viremia and/or Viruria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 071A; Study No B102
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-12

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Immunotherapy; Drug Evaluation; Cytomegalovirus Infections; Antibodies, Monoclonal
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; AIDS-Related Opportunistic Infections | interventions — sevirumab

INTERVENTIONS:
Drug: Sevirumab

SUMMARY:
To determine the safety, tolerance, and potential in vivo antiviral effects of five dosage levels and a dose to be determined of human anti-cytomegalovirus (CMV) monoclonal antibody (SDZ MSL-109; formerly SDZ 89-109) when administered once every 2 weeks for a total of 12 doses to patients with either AIDS or eligible AIDS-related complex (ARC) and with culture proven evidence of CMV viremia and/or viruria. Sandoglobulin will be employed as a comparative control.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* Acyclovir.
* Experimental maintenance or prophylactic therapy with an approved therapeutic agent for a non-viral opportunistic infection.
* Trimethoprim / sulfamethoxazole (TMP / SMX).
* Pyrimethamine / sulfadoxine.
* Inhaled pentamidine.
* Amphotericin B.
* Ketoconazole.
* Flucytosine (5-FC).
* Antituberculosis therapy.
* Recombinant human erythropoietin.
* Recombinant granulocyte-macrophage colony-stimulating factor (GM-CSF).
* Recombinant human interferon alfa 2 for AIDS-related Kaposi's sarcoma.

Patients must have:

* AIDS or be HIV positive with CD4 lymphocyte counts below 200 cells/mm3 and be receiving prophylaxis for Pneumocystis carinii pneumonia (PCP) (with or without prophylaxis for another opportunistic infection), but have no prior medical history of an opportunistic infection.
* Expected survival of = or > 6 months.
* Willingness and ability to give written informed consent.
* A copy of the signed and witnessed consent form must be maintained with the investigator's study files.
* Positive culture results documenting the presence of cytomegalovirus (CMV) viremia and/or viruria.
* Seropositive for the presence of circulating anti-CMV immunoglobulin.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Significant pulmonary dysfunction.
* Uncontrolled or unstable diabetes.
* Significant cardiovascular disease including uncontrolled hypertension, congestive heart failure, cardiac arrhythmia, angina pectoris, or a history of myocardial infarction within one year of entry into the study.
* Coagulation or hemorrhagic disorders.
* Any active severe opportunistic infection.

Concurrent Medication:

Excluded:

* Therapy with ganciclovir (DHPG) or phosphonoformate (PFA) or other experimental anti-cytomegalovirus therapy except as stipulated in this protocol.
* Any other experimental antiviral therapy.
* Biologicals including immunoglobulin therapy (except those patients randomized to receive Sandoglobulin as specified in this protocol).

Patients with the following are excluded:

* Any significant organ system dysfunction as described in Exclusion co-existing conditions.
* Previous history of or evidence of idiopathic thrombocytopenia purpura, agammaglobulinemia, or hypogammaglobulinemia.
* Any other severe concomitant clinical condition.
* Documented, active cytomegalovirus (CMV) disease (tissue or organ invasion/dysfunction) at baseline. To this end, baseline indirect funduscopy (to detect and exclude patients with peripheral CMV retinitis) will be performed.

Prior Medication:

Excluded within 2 weeks of study entry:

* Therapy with ganciclovir (DHPG) or phosphonoformate (PFA) or other experimental anti-cytomegalovirus therapy except as stipulated in this protocol.
* Any other experimental antiviral therapy.
* Biologicals including immunoglobulin therapy (except those patients randomized to receive Sandoglobulin as specified in this protocol).
* Excluded:
* Prior treatment with monoclonal antibodies derived from any animal species.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ TX Galveston Med Branch, Galveston, Texas